CLINICAL TRIAL: NCT05745259
Title: Thrombolysis Treated by TNK-tPA in Acute Ischemic Stroke Patients: a Multi-center, Block Randomized, Positive Drug Parallel Control and Non-inferior Phase Ⅲ Trial, 3T Stroke-Ⅲ
Brief Title: Thrombolysis Treated With TNK-tPA in Acute Ischemic Stroke Patients （3T Stroke-Ⅲ）
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Beijing Tiantan Hospital (Other)
Collaborators: Jiangsu FENG HUA Biotech Pharmaceutical Co., Ltd (Unknown); The Place Pharmaceutical(Jiangsu) Co., Ltd (Unknown)
Responsible Party: Principal Investigator, Yongjun Wang, President of Beijing Tiantan Hospital, Capital Medical University, Director of Neurology Center, Beijing Tiantan Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PR-FHSW-2022001F
Record Dates: First submitted 2023-02-16; First posted 2023-02-27 (Actual); Last update posted 2023-02-27 (Actual); Status verified 2023-02

CONDITIONS: Acute Ischemic Stroke
Keywords: TNK-tPA, rt-PA, Acute stroke, phase Ⅲ trial
MeSH Terms: conditions — Ischemic Stroke; Stroke | interventions — Tissue Plasminogen Activator; Tenecteplase; TNK-tissue plasminogen activator

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Alteplase (Active Comparator): Patients will receive intravenous Alteplase at the standard licensed dose of 0.9 mg/kg up to a maximum of 90mg, 10% as bolus and the remainder over 1 hour.
  Interventions: Drug: Alteplase
- Tenecteplase (Experimental): Patients will receive intravenous Tenecteplase, 0.25mg/kg, maximum 25mg, administered as a bolus over 5~10 seconds
  Interventions: Drug: Tenecteplase

INTERVENTIONS:
Drug: Alteplase — Alteplase 0.9mg/kg are being used.
  Other Names: rt-PA
  Arms: Alteplase
Drug: Tenecteplase — Tenecteplase 0.25mg/kg are being used.
  Other Names: TNK-tPA
  Arms: Tenecteplase

SUMMARY:
The trial is prospective, randomized, open-label, blinded endpoint (PROBE) design. Patients with acute ischemic stroke, who are eligible for standard intravenous thrombolysis within 4.5 hours of stroke onset will be randomized 1:1 to 0.25mg/kg or 0.9 mg/kg alteplase before all participants undergo endovascular thrombectomy.

DETAILED DESCRIPTION:
The study will be a multi-center, prospective, randomized, open- label, blinded endpoint (PROBE), controlled phase 3 trial (2 arm with 1:1 randomization) in ischemic stroke patients. Imagine is performed with CT or MRI acutely with imaging follow-up at 24-36 hours. The sample size is 1630.

ELIGIBILITY:
Inclusion Criteria:

* 18≤Age≤80 years old;
* The clinical diagnosis was Acute ischemic stroke The time from onset to treatment was < 4.5h; The time at which symptoms begin is defined as "the time at which they finally appear normal";
* MRS before onset was ≤1 points;
* Baseline NIHSS (at the time of randomization) should be ≥5 and ≤25 points;
* Informed consent from the patient or surrogate.

Exclusion Criteria:

* Intracranial hemorrhage identified by CT or MRI (CMBs detected by SWI is not counted);
* Massive anterior cerebral infarction identified by CT or MRI (ASPECT < 6 or lesions larger than one third of the territory of the middle cerebral artery or with a volume larger than 70mL)
* Patients planning to receive endovascular therapy
* A history of severe CNS damage (such as aneurysm or arteriovenous malformation, craniocerebral trauma, intracranial or spinal cord surgery)
* Onset with seizures, and the paralysis was suspected to be related to Todd paralysis.
* Administration of heparin within 48 hours preceding the onset of stroke with a baseline APTT exceeding the upper limit of the normal range.
* Oral anticoagulant (such as warfarin) treatment with baseline INR>1.7 or PT>15 s;
* Administration of thrombin inhibitors or factor Xa inhibitors within 48 hours preceding the onset of stroke with abnormal coagulation parameters or platelet count;
* BP couldn't be controlled with aggressive treatment. Uncontrolled hypertension was defined as systolic blood pressure >185 mmHg or diastolic blood pressure >110 mmHg, measured for three times every 10 minutes.
* Platelet count of less than 100×109/ L;
* Blood glucose <50 mg/dl (<2.8 mmol/L) or >400 mg/dl (22.22 mmol/L);
* History of intracranial hemorrhage or active hemorrhagic disease. (Such as gastrointestinal, urinary tract or retinal bleeding)
* Tumors with an increased risk of bleeding.
* Prolonged or traumatic cardiopulmonary resuscitation (>2 min), delivery within the last 10 days or recent puncture of non-compression vessels such as subclavian vein or jugular vein
* Acute pancreatitis or severe liver disease, including liver failure, cirrhosis, portal hypertension, esophageal varicose veins, and active hepatitis;
* Aortic arch dissection;
* Major surgery or severe trauma in the past 2 weeks;
* Subjects had serious, fatal, or disabling disease with an expected survival of less than 3 months;
* Unable to complete neurological assessment and follow-up visits because of dementia or mental illness;
* Pregnant women, lactating women, or have positive pregnancy test;
* Allergy to tenecteplase or alteplase or their components;
* Participation in other clinical trials within 3 months prior to screening;
* Unsuitable to involve in this study or would result in increased risk, as judged by the investigators.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1630 (Estimated)
Dates: Start 2022-10-26 (Actual); Primary Completion 2023-11-04 (Estimated); Study Completion 2024-03-29 (Estimated)

PRIMARY OUTCOMES:
Modified Rankin Scale(mRS) | 90±7 days
  Proportion of subjects with mRS scores of (0-1) at 90±7 days.

SECONDARY OUTCOMES:
National Institutes of Health Stroke Scale (NIHSS) | 24±2 hours
  NIHSS score at 24±2 hours.
National Institutes of Health Stroke Scale (NIHSS) | 7±2days or discharge
  Proportion of subjects with ≥ 4 point reduction in NIHSS or reaching 0-1 at 7 ± 2 days or before discharge (whichever occurs first)
Modified Rankin Scale(mRS) | 90±7 days
  Proportion of subjects with mRS scores of (0-2) at 90±7 days.
Modified Rankin Scale(mRS) | 90±7 days
  mRS scores at 90±7 days.
The new vascular events | 90±7 days
  Incidence of the new vascular events, ischemic stroke, hemorrhagic stroke, myocardial infarction and cardio-cerebral revascularization at 90±7 days. (including: carotid endarterectomy, intracranial and extracranial artery interventional therapy, intracranial and extracranial artery bypass surgery, coronary interventional or bypass therapy)
EQ-5D | 90±7 days
  EQ-5D scores at 90±7 days.

OTHER OUTCOMES:
Symptomatic intracranial hemorrhage(sICH) | 24~36 hours post treatment
  Incidence of symptomatic intracranial hemorrhage (sICH) within 24~36 hours.( According to ECASS Ⅲ and SITS-MOST)
Parenchymal hematoma intracranial hemorrhage (type PH2, SITS-MOST) | 24~36 hours post treatment
  Incidence of intracranial hemorrhage (type PH2, SITS-MOST) within 24~36 hours.
Any intracranial hemorrhage | 24~36 hours post treatment
  Incidence of any intracranial hemorrhage within 24~36 hours.
Systematic bleeding | 36 hours
  Incidence of Systematic bleeding within 36 hours. (defined by GUSTO)
Deaths | 90±7 days
  Vascular mortality at 90±7 days (mainly due to stroke, myocardial infarction or pulmonary embolism)
Deaths | 90±7 days
  Mortality due to any cause at 90±7days.
SAEs | 90±7 days
  Incidence of severe adverse events(SAEs) at 90±7 days.
AEs | 90±7 days
  Incidence of adverse events(AEs) at 90±7 days.

CONTACTS AND LOCATIONS:
Overall Officials: Shuya Li, Study Director — IRB of Beijing Tiantan Hospital,Capital Medical University
Locations (63):
- China (63):
  - Xuancheng People's Hospital, Xuancheng, Anhui
  - Beijing Tiantan Hospital, Capital Medical University Beijing, Beijing, Beijing Municipality
  - Xuanwu Hospital Capital Medical University, Beijing, Beijing Municipality
  - Three Gorges Hospital Affiliated to Chongqing University, Chongqing, Chongqing Municipality
  - Quanzhou First Hospital, Quanzhou, Fujian
  - Lanzhou University First Hospital, Lanzhou, Gansu
  - The Third People's Hospital of Huizhou, Huizhou, Guangdong
  - Yuebei People's Hospital, Shaoguan, Guangdong
  - The First People's Hospital of Yulin, Yulin, Guangxi
  - Handan Central Hospital, Handan, Hebei
  - Hengshui people's Hospital (Harrison International Peace Hospital), Hengshui, Hebei
  - Tangshan Workers' Hospital, Tangshan, Hebei
  - Daqing Oilfield General Hospital, Daqing, Heilongjiang
  - Daqing People's Hospital, Daqing, Heilongjiang
  - Anyang People's Hospital, Anyang, Henan
  - Jiaozuo People's Hospital, Jiaozuo, Henan
  - Nanyang South Stone Hospital, Nanyang, Henan
  - Pingmei Shenma medical group general hospital, Pingdingshan, Henan
  - Xinxiang Central Hospital, Xinxiang, Henan
  - Zhoukou Downtown Hospital, Zhoukou, Henan
  - The First People's Hospital of Jingzhou, Jingzhou, Hubei
  - Baogang Hospital of Inner Monglia, Baotou, Inner Monglia
  - Baotou Central Hospital, Baotou, Inner Mongolia
  - Keshenketengqi Mongolian Medicine Hospital, Chifeng, Inner Mongolia
  - The Second Affiliated Hospital of Suzhou Medical University, Suzhou, Jiangsu
  - Taizhou People's Hospital, Taizhou, Jiangsu
  - Xuzhou Central Hospital, Xuzhou, Jiangsu
  - Xuzhou Mining Group General Hospital, Xuzhou, Jiangsu
  - The Affiliated Hospital of Xuhzou Meidcal University, Xuzhou, Jiangsu
  - The First Hospital of Jilin University, Changchun, Jilin
  - Jilin Guowen Hospital, Siping, Jilin
  - Siping Central People's Hospital, Siping, Jilin
  - Tonghua Central Hospital, Tonghua, Jilin
  - Meihekou Central Hospital, Tonghua, Jilin
  - Beipiao Central Hospital, Beipiao, Liaoning
  - Dalian Central Hospital, Dalian, Liaoning
  - Fushun Mining Bureau General Hospital, Fushun, Liaoning
  - Liaoning Health Industry Group Fuxin Mine General Hospital, Fuxin, Liaoning
  - The First Affiliated Hospital of Jinzhou Medical University, Jinzhou, Liaoning
  - Affiliated Central Hospital of Shenyang Medical College, Shenyang, Liaoning
  - Air Force Hospital of Northern War Zone,PLA, Shenyang, Liaoning
  - General Hospital of Northern War Zone,PLA, Shenyang, Liaoning
  - The First Affiliated Hospital of China Medical University, Shenyang, Liaoning
  - The First People's Hospital of Shenyang, Shenyang, Liaoning
  - General Hospital of Ningxia Medical University Cardio-cerebral Vascular Disease Hospital, Yinchuan, Ningxia
  - The First People's Hospital of Yinchuan, Yinchuan, Ningxia
  - Dezhou Hospital of Shandong University Qilu Hospital (Dezhou People's Hospital), Dezhou, Shandong
  - Jinan People's Hospital, Jinan, Shandong
  - Qilu Hospital of Shandong University, Jinan, Shandong
  - Liaocheng People's Hospital, Liaocheng, Shandong
  - Linyi Hospital of Traditional Chinese Medicine, Linyi, Shandong
  - Linyi People's Hospital, Linyi, Shandong
  - The First People's Hospital of Tancheng County, Linyi, Shandong
  - Taian Central Hospital (Tai 'an Central Hospital of Qingdao University, Tai 'an Medical and Nursing Center), Taian, Shandong
  - Tengzhou Central Hospital, Tengzhou, Shandong
  - Weifang Hospital of Traditional Chinese Medicine, Weifang, Shandong
  - Yantai Yuhangding Hospital, Yantai, Shandong
  - Sinopharm Coal Mine General Hospital, Datong, Shanxi
  - Linfen Central Hospital, Linfen, Shanxi
  - Linfen People's Hospital, Linfen, Shanxi
  - Shanxi Cardiovascular Disease Hospital, Taiyuan, Shanxi
  - Dazhu County People's Hospital, Dazhu, Sichuan
  - Mianyang Central Hospital, Mianyang, Sichuan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Guidelines Editing Group of Chinese Stroke Society, Guidelines for the Diagnosis and Treatment of High-risk Non-Disabling Ischemic Cerebrovascular Events, Chinese Journal of Stroke, June 2016, 11 (6), p481-491.
- [Background] Chinese Journal of Circulation, China Cardiovascular Disease Report 2015.
- [Background] CAST: randomised placebo-controlled trial of early aspirin use in 20,000 patients with acute ischaemic stroke. CAST (Chinese Acute Stroke Trial) Collaborative Group. Lancet. 1997 Jun 7;349(9066):1641-9. PMID 9186381
- [Background] Hao Zilong, Liu Ming, Li Wei, et al. Stroke registration method and basic characteristics and functional outcomes of 3123 patients in Chengdu [J]. Chinese Journal of Neurology, 2011,12 (44) : 826-831.
- [Background] Wang Z, Li J, Wang C, Yao X, Zhao X, Wang Y, Li H, Liu G, Wang A, Wang Y. Gender differences in 1-year clinical characteristics and outcomes after stroke: results from the China National Stroke Registry. PLoS One. 2013;8(2):e56459. doi: 10.1371/journal.pone.0056459. Epub 2013 Feb 13. PMID 23418571
- [Background] Wei JW, Heeley EL, Wang JG, Huang Y, Wong LK, Li Z, Heritier S, Arima H, Anderson CS; ChinaQUEST Investigators. Comparison of recovery patterns and prognostic indicators for ischemic and hemorrhagic stroke in China: the ChinaQUEST (QUality Evaluation of Stroke Care and Treatment) Registry study. Stroke. 2010 Sep;41(9):1877-83. doi: 10.1161/STROKEAHA.110.586909. Epub 2010 Jul 22. PMID 20651267
- [Background] Bandera E, Botteri M, Minelli C, Sutton A, Abrams KR, Latronico N. Cerebral blood flow threshold of ischemic penumbra and infarct core in acute ischemic stroke: a systematic review. Stroke. 2006 May;37(5):1334-9. doi: 10.1161/01.STR.0000217418.29609.22. Epub 2006 Mar 30. PMID 16574919
- [Background] Donnan GA, Baron JC, Ma H, Davis SM. Penumbral selection of patients for trials of acute stroke therapy. Lancet Neurol. 2009 Mar;8(3):261-9. doi: 10.1016/S1474-4422(09)70041-9. PMID 19233036
- [Background] Haley EC Jr, Thompson JL, Grotta JC, Lyden PD, Hemmen TG, Brown DL, Fanale C, Libman R, Kwiatkowski TG, Llinas RH, Levine SR, Johnston KC, Buchsbaum R, Levy G, Levin B; Tenecteplase in Stroke Investigators. Phase IIB/III trial of tenecteplase in acute ischemic stroke: results of a prematurely terminated randomized clinical trial. Stroke. 2010 Apr;41(4):707-11. doi: 10.1161/STROKEAHA.109.572040. Epub 2010 Feb 25. PMID 20185783
- [Background] Parsons M, Spratt N, Bivard A, Campbell B, Chung K, Miteff F, O'Brien B, Bladin C, McElduff P, Allen C, Bateman G, Donnan G, Davis S, Levi C. A randomized trial of tenecteplase versus alteplase for acute ischemic stroke. N Engl J Med. 2012 Mar 22;366(12):1099-107. doi: 10.1056/NEJMoa1109842. PMID 22435369
- [Background] Huang X, Cheripelli BK, Lloyd SM, Kalladka D, Moreton FC, Siddiqui A, Ford I, Muir KW. Alteplase versus tenecteplase for thrombolysis after ischaemic stroke (ATTEST): a phase 2, randomised, open-label, blinded endpoint study. Lancet Neurol. 2015 Apr;14(4):368-76. doi: 10.1016/S1474-4422(15)70017-7. Epub 2015 Feb 26. PMID 25726502
- [Background] Logallo N, Novotny V, Assmus J, Kvistad CE, Alteheld L, Ronning OM, Thommessen B, Amthor KF, Ihle-Hansen H, Kurz M, Tobro H, Kaur K, Stankiewicz M, Carlsson M, Morsund A, Idicula T, Aamodt AH, Lund C, Naess H, Waje-Andreassen U, Thomassen L. Tenecteplase versus alteplase for management of acute ischaemic stroke (NOR-TEST): a phase 3, randomised, open-label, blinded endpoint trial. Lancet Neurol. 2017 Oct;16(10):781-788. doi: 10.1016/S1474-4422(17)30253-3. Epub 2017 Aug 2. PMID 28780236
- [Background] Campbell BCV, Mitchell PJ, Churilov L, Yassi N, Kleinig TJ, Dowling RJ, Yan B, Bush SJ, Dewey HM, Thijs V, Scroop R, Simpson M, Brooks M, Asadi H, Wu TY, Shah DG, Wijeratne T, Ang T, Miteff F, Levi CR, Rodrigues E, Zhao H, Salvaris P, Garcia-Esperon C, Bailey P, Rice H, de Villiers L, Brown H, Redmond K, Leggett D, Fink JN, Collecutt W, Wong AA, Muller C, Coulthard A, Mitchell K, Clouston J, Mahady K, Field D, Ma H, Phan TG, Chong W, Chandra RV, Slater LA, Krause M, Harrington TJ, Faulder KC, Steinfort BS, Bladin CF, Sharma G, Desmond PM, Parsons MW, Donnan GA, Davis SM; EXTEND-IA TNK Investigators. Tenecteplase versus Alteplase before Thrombectomy for Ischemic Stroke. N Engl J Med. 2018 Apr 26;378(17):1573-1582. doi: 10.1056/NEJMoa1716405. PMID 29694815
- [Background] Emberson J, Lees KR, Lyden P, Blackwell L, Albers G, Bluhmki E, Brott T, Cohen G, Davis S, Donnan G, Grotta J, Howard G, Kaste M, Koga M, von Kummer R, Lansberg M, Lindley RI, Murray G, Olivot JM, Parsons M, Tilley B, Toni D, Toyoda K, Wahlgren N, Wardlaw J, Whiteley W, del Zoppo GJ, Baigent C, Sandercock P, Hacke W; Stroke Thrombolysis Trialists' Collaborative Group. Effect of treatment delay, age, and stroke severity on the effects of intravenous thrombolysis with alteplase for acute ischaemic stroke: a meta-analysis of individual patient data from randomised trials. Lancet. 2014 Nov 29;384(9958):1929-35. doi: 10.1016/S0140-6736(14)60584-5. Epub 2014 Aug 5. PMID 25106063
- [Background] National Institute of Neurological Disorders and Stroke rt-PA Stroke Study Group. Tissue plasminogen activator for acute ischemic stroke. N Engl J Med. 1995 Dec 14;333(24):1581-7. doi: 10.1056/NEJM199512143332401. PMID 7477192
- [Background] Hacke W, Kaste M, Fieschi C, von Kummer R, Davalos A, Meier D, Larrue V, Bluhmki E, Davis S, Donnan G, Schneider D, Diez-Tejedor E, Trouillas P. Randomised double-blind placebo-controlled trial of thrombolytic therapy with intravenous alteplase in acute ischaemic stroke (ECASS II). Second European-Australasian Acute Stroke Study Investigators. Lancet. 1998 Oct 17;352(9136):1245-51. doi: 10.1016/s0140-6736(98)08020-9. PMID 9788453
- [Background] Clark WM, Wissman S, Albers GW, Jhamandas JH, Madden KP, Hamilton S. Recombinant tissue-type plasminogen activator (Alteplase) for ischemic stroke 3 to 5 hours after symptom onset. The ATLANTIS Study: a randomized controlled trial. Alteplase Thrombolysis for Acute Noninterventional Therapy in Ischemic Stroke. JAMA. 1999 Dec 1;282(21):2019-26. doi: 10.1001/jama.282.21.2019. PMID 10591384
- [Background] Zheng H, Yang Y, Chen H, Li C, Chen Y, Shi FD, Yang L, Cui X, Lu Z, Liang Y, Cui S, Xu A, Wu Y, Sun Y, Wang Y. Thrombolysis with alteplase 3-4.5 hours after acute ischaemic stroke: the first multicentre, phase III trial in China. Stroke Vasc Neurol. 2020 Sep;5(3):285-290. doi: 10.1136/svn-2020-000337. Epub 2020 May 28. PMID 32467323
- [Background] Standards and procedures for rapid reporting of safety data during drug clinical trials